CLINICAL TRIAL: NCT07168330
Title: Clinical and Radiological Evaluation in Patients With Total Ankle Replacement
Brief Title: Clinical and Radiological Evaluation of Total Ankle Replacement (ProtesiTT)
Acronym: ProtesiTT
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: ProtesiTT
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Ankle replacement — Total ankle arthroplasty

SUMMARY:
Numerous studies reported the efficacy of new third-generation of total ankle arthroplasties for the treatment of advanced ankle osteoarthritis and clinical results are comparable to ankle arthrodesis. The improvement in knowledge of ankle joint biomechanics, instrumentation, surgical approach may led to even higher clinical results in comparison to arthrodesis.

Many of the studies reporting the results of ankle replacement are provided by surgeons involved at least in the initial design of the implant. Thus, familiarity with the system can be a potential bias affecting outcomes and orthopedic surgeons may find difficulties in reproducing the results.

In this study, we will assess the clinical and radiological outcomes in patients who underwent this procedure performed by non-designer surgeons

DETAILED DESCRIPTION:
Patients who underwent total ankle replacement will be unrolled in this study. Clinical assessment is collected pre- and post-operatively with minimum follow-up of 12 months from each patients using the American Orthopedic Foot and Ankle (AOFAS) score, the Foot Function Index and the visual analogue scale (VAS) for pain.

Weightbearing anteriorposterior and lateral radiographs of the ankle are collected pre-operatively and at the last follow-up for all of the patients and independently evaluated by an orthopedic surgeon.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with ankle replacement for osteoarthritis
* The patient is willing and able to complete scheduled follow-up evaluations questionnaires and radiographic examination as described in the Informed Consent

Exclusion Criteria:

* patients without radiographic follow-up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with ankle replacement for osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
survivorship | 10 years
  Survival of the implants after 10 years which is based on removal of the components and will be assessed using the Kaplan Meier Method

SECONDARY OUTCOMES:
angle a | 10 years
  radiographic outcome
angle b | 10 years
  radiographic Outcome
angle y | 10 years
  radiographic Outcome
offset ratio | 10 years
  radiographic Outcome
AOFAS score | 10 years
  Clinical Outcome; American Orthopaedic Foot and Ankle Society: from 0 (severe) to 100 (not severe)
Foot function Index | 10 years
  Clinical outcome; from 0 (not severe) to 10 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Bianchi, MD, Principal Investigator — IRCCS Galeazzi, Foot and Ankle Department
Locations (1):
- IRCCS Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided